CLINICAL TRIAL: NCT03329131
Title: Evaluation of Cryotherapy and TRPA1 Receptors in Chemotherapy Induced Neuropathy
Brief Title: Breast/Evaluation of Cryotherapy and TRPA1 Receptors in Chemotherapy Induced Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Virginia G. Kaklamani, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTMS #17-0033; HSC20170535H (Other: UT Health San Antonio)
Record Dates: First submitted 2017-09-27; First posted 2017-11-01 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Neuropathies
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cryotherapy (Experimental): Each patient will receive cryotherapy administered during each neurotoxic chemotherapy agent infused treatments by Elasto gel™ Hypothermia gloves and socks. Patients will wear the glove and sock for 15 minutes prior to treatment start and 15 minutes following treatment completion, for a total of 30 minutes.
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Cryotherapy — An Elasto gel™ frozen (4°C) glove and sock
  Other Names: Cold therapy; Elasto gel™

SUMMARY:
To determine rate and severity of chemotherapy induced neuropathy in extremities treated with cold gloves and socks versus control extremities

DETAILED DESCRIPTION:
This is a therapeutic study investigating the use of cryotherapy in the prevention of chemotherapy-induced peripheral neuropathy (CIPN) and associated nail toxicities. The therapeutic intervention will involve patients wearing an Elasto-Gel cold glove and sock on one hand and one foot (both on the right side or both on the left side). The patients will wear the glove and sock during each infusion of taxane chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of early stage breast cancer (stage I-III).
* Planned to receive treatment with either adjuvant or neo-adjuvant taxane-based chemotherapy.
* Age > 18 years. There is no upper age limit for participation in this study.
* Patients may have received any of the following therapies: surgery, chemotherapy, hormones, biologics, or radiation.
* Prior chemotherapies are permitted, except with prior treatments with taxanes, vinca alcaloids, gemcitabine, eribulin, ixabepilone, platinum drugs)
* All patients will have given signed, informed consent prior to registration
* Patients must have a performance status of ECOG 0 or 1.

Exclusion Criteria

* Patients must not have received any prior taxane or platinum based chemotherapy.
* Patients must not have a history of peripheral neuropathy (regardless of cause).
* Patient must not have a history of Raynaud's disease.
* Patients with partial or complete limb amputations.
* Known hypersensitivity to cold
* Patient cannot be on the following medications: GABA analogues (such as Neurontin, lyrica), tricyclic antidepressants (such as amitriptyline or nortriptyline)
* As judged by the investigator, severe uncontrolled concurrent medical conditions, psychiatric illness or social condition that would limit compliance with study requirements.
* Evidence of any significant clinical disorder or laboratory finding that makes it undesirable for the subject to participant in the clinical trial
* Must not be pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health Cancer Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryotherapy
Started | 12
Completed | 8
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: This is a therapeutic study investigating the use of cryotherapy in the prevention of chemotherapy-induced peripheral neuropathy (CIPN) and associated nail toxicities. The therapeutic intervention will involve patients wearing an Elasto-Gel cold glove and wrap on one hand and one foot (both on the right side or both on the left side). The patients will wear the glove and wrap during each infusion of taxane chemotherapy.
Arm/Group | Cryotherapy
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Peripheral Neuropathy During Taxane Chemotherapy
Description: A Visual analog scale (VAS) was used to assess change in pain after using a mustard oil challenge from pre- to post-infusion and the results reported as an average. The Visual Analogue Scale (VAS) is a tool that measures pain intensity by asking a patient to mark a point on a 100 mm line that represents their current pain level. The line has two endpoints, with 0mm representing "no pain" and 100mm representing "pain as bad as it could possibly be". The patient's score is determined by measuring the distance in millimeters from the left end of the line to the point they mark. A higher score indicates greater pain intensity.
Time Frame: Change from baseline to 6 months post chemo (up to 14 months)
Population: Only 7 of the subjects were evaluable, and not all data from all time points was available due to suspension of research activities during the pandemic
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cryotherapy
Number analyzed (Participants) | 7
score on a scale | 7.28 [0 to 29]

2. Primary Outcome: Evaluate Safety of Cryotherapy Use
Description: Number of Adverse events Grade 3 or higher attributed to the use of Cryotherapy according to the National Cancer Institute - Common Terminology Criteria for Adverse Events NCI-CTCAE v 4.03 Assessment for peripheral neuropathy and nail changes
Time Frame: Baseline to 6 months post Cryotherapy (up to 14 months)
Population: Only 8 of the subjects were evaluable for adverse events of Grade 3 or higher, and not all data from all time points was available due to suspension of research activities during the pandemic
Measure: Number; unit: Number of Adverse Events
Arm/Group | Cryotherapy
Number analyzed (Participants) | 8
Number of Adverse Events | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to 6 months post chemotherapy (variable depending on number of cycles of chemotherapy administered up to 14 months)
Description: For this study, all adverse events will be documented starting with the first use of the cold therapy device and ending 30 days after the last dose use of the cold therapy device, regardless of the length of time the device was used.
Arm/Group | Cryotherapy
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy (N=12)
Peripheral neuropathy (Nervous system disorders) | 3 (7) — Related to chemotherapy, not cryotherapy
Fever (General disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Fatigue (General disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Myalgia (Nervous system disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Nausea (Gastrointestinal disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Rash on hands (Skin and subcutaneous tissue disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Bone pain (General disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Dry skin on feet (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (General disorders) | 1 (1) — Related to chemotherapy, not cryotherapy
Nail bed changes (Skin and subcutaneous tissue disorders) | 1 (1) — Related to Chemotherapy not cryotherapy
Rectal bleeding (Gastrointestinal disorders) | 1 (1) — Rectal bleeding with bowel movement, not related to cryotherapy
Nail bed loss (Skin and subcutaneous tissue disorders) | 1 (1) — Related to chemotherapy, not cryotherapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03329131/Prot_SAP_000.pdf